CLINICAL TRIAL: NCT05007756
Title: A Phase 0 Platform Study Exploring the Use of Challenge Agents in Healthy Volunteers or Participants With a Disease of Interest
Brief Title: A Study Exploring the Use of Challenge Agents in Healthy Volunteers or Participants With a Disease of Interest
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR109034; NOPRODPCNAP0002 (Other: Janssen Research & Development, LLC); PLATFORMPCNAP0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-07-12; First posted 2021-08-16 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultraviolet B (UVB) Challenge (Experimental): Participants will receive UVB (various doses) for minimal erythema dose (MED) assessment at baseline following which there will be washout period. Participants will then receive a single dose of UVB challenge dermally through Lumera Phototherapy System on Day 1, twice (2*) the MED at the challenge site with no UVB exposure at the contralateral control site.
  Interventions: Radiation: UVB Challenge

INTERVENTIONS:
Radiation: UVB Challenge — UVB challenge will be administered dermally through Lumera Phototherapy System.

SUMMARY:
The purpose of this study is to characterize the biological response in vivo to challenge agents (vaccines, antigen, drug, or mechanical challenges); to assess the safety and tolerability of the challenge agent and to characterize the immune response in skin elicited in vivo in healthy volunteers using an ultraviolet B (UVB) challenge.

ELIGIBILITY:
Inclusion Criteria:

* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-HCG]) at screening and a negative urine pregnancy test prior to study intervention administration on Day -4
* Must have Fitzpatrick skin type II or III (10 participants) or type IV or higher (2 participants)
* Otherwise healthy on the basis of physical examination, medical history, and vital signs, and, if required by the applicable Intervention Specific Appendix (ISA), a 12-lead Electrocardiography (ECG) performed at screening. Any abnormalities must be considered not clinically significant or consistent with the underlying illness in the study population and this determination must be recorded
* Otherwise healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Must be a non-smoker (not smoked for at least 6 months prior to screening) and has not used nicotine-containing products (example, nicotine patch) for 3 months prior to screening

Exclusion Criteria:

* Has a history of dysplastic melanocytic nevi or skin cancer
* Known hypersensitivity, intolerance to UV/sunlight exposure, or any condition associated with photosensitivity
* Has Fitzpatrick skin type I, as determined by the investigator. A person with Fitzpatrick skin type I typically has unexposed skin that is bright white with frequent freckling, has blue/green eyes, and is of Northern European/British descent. They typically burn, peel, and don't tan in response to ultraviolet B (UVB)
* Has a history of chronic skin conditions, such as vitiligo, psoriasis, rosacea, severe eczema, or atopic dermatitis, and/or severe acne that would complicate or preclude evaluation of the minimal erythema dose (MED) testing and UVB challenge sites
* Has used topical antibiotics or topical corticosteroids within 1 month prior to study intervention administration and/or has a history of extensive and prolonged use (greater than [>] 3 months) of topical antibiotics or topical corticosteroids

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Changes in Gene Expression as Measured by Counts of Transcript per Million Reads | Up to Week 6
  Changes in gene expression as measured by counts of transcript per million reads in control versus challenged tissue will be reported.
Changes in Gene Set Variation Analysis Enrichment Score | Up to Week 6
  Changes in gene set variation analysis (GSVA) enrichment score control versus challenged tissue will be reported. The GSVA score is a measurement of changes in a set of genes between 2 sample sets (example, control versus test).
Changes in Cell Count as Measured by Fluorescence Intensity | Up to Week 6
  Changes in cell count as measured by fluorescence intensity via immunohistochemistry (IHC) in control versus challenged tissue will be reported.
Changes in Protein Expression as Measured by Fluorescence Intensity | Up to Week 6
  Changes in protein expression as measured by fluorescence intensity via IHC in control versus challenged tissue will be reported.
Changes in Gene Expression as Measured by Fluorescence Intensity | Up to Week 6
  Changes in gene expression as measured by fluorescence intensity via IHC in control versus challenged tissue will be reported.
Changes in the Levels of Proteins and Phosphoproteins | Up to Week 6
  Changes in the levels of proteins and phosphoproteins which are relevant to inflammatory pathways thought to be activated by ultraviolet B (UVB) exposure (example, Type 1 interferons pathways) measured by enzyme-linked immunoassay (ELISA) in control versus challenged tissue lysates, will be reported.
Fold Changes in the Mean Differences of the Levels of Proteins and Phosphoproteins | Up to Week 6
  Fold changes in the mean differences of the levels of the proteins and phosphoproteins which are relevant to inflammatory pathways thought to be activated by UVB exposure (example, type 1 interferons pathways) measured by ELISA in control versus challenged tissue lysates, will be reported.
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Week 6
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Treatment-emergent Serious Adverse Events (SAEs). | Up to Week 6
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent SAEs are defined as serious events between administration of study drug and after the last dose that were absent before treatment or that worsen relative to pretreatment state.
Number of Participants with TEAEs by Medical Dictionary for Regulatory Activities (MedDRA) System-organ Class (SOC) with a Frequency Threshold of at Least 2 Participants per Intervention Cohort | Up to Week 6
  Number of participants with TEAEs by MedDRA SOC with a frequency threshold of at least 2 participants per intervention cohort will be reported. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.

SECONDARY OUTCOMES:
Standard Deviation of Changes in Gene Expression as Measured by Counts of Transcript per Million Reads | Up to Week 6
  Standard deviation of changes in gene expression as measured by counts of transcript per million reads in control versus challenged tissue will be reported.
Standard Deviation of Changes in GSVA Enrichment Score | Up to Week 6
  Standard deviation of changes in GSVA enrichment score will be reported. The GSVA score is a measurement of changes in a set of genes between 2 sample sets (example, control versus test).
Standard Deviation of Changes in Cell Count as Measured by Fluorescence Intensity | Up to Week 6
  Standard deviation of changes in cell count as measured by fluorescence intensity via IHC in control versus challenged tissue will be reported.
Standard Deviation of Changes in Protein Expression as Measured by Fluorescence Intensity | Up to Week 6
  Standard deviation of changes in protein expression as measured by fluorescence intensity via immunohistochemistry (IHC) in control versus challenged tissue will be reported.
Standard Deviation of Changes in Gene Expression as Measured by Fluorescence Intensity | Up to Week 6
  Standard deviation of changes in gene expression as measured by fluorescence intensity via IHC in control versus challenged tissue will be reported.
Standard Deviation of Changes in Phosphoproteins and Other Proteins | Up to Week 6
  Standard deviation of changes in phosphoproteins and other proteins in tissue lysate in control versus challenged tissue will be reported.
Standard Deviation of Fold Changes of Means of Phosphoproteins and Other Proteins | Up to Week 6
  Standard deviation of fold changes of means of phosphoproteins and other proteins in control versus challenged tissue will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency